CLINICAL TRIAL: NCT04748770
Title: Access to Kidney Transplant of Obese Patients Beginning Dialysis
Acronym: Transplantob
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2021_843_0016
Record Dates: First submitted 2021-02-09; First posted 2021-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Kidney Transplant Access; Obese Patients; Dialysis; Comorbidities
Keywords: Kidney transplant access; obese patients; dialysis; comorbidities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with BMI≥30 kg/m2
- patients with 25≤BMI≤30 kg/m2

SUMMARY:
Obesity is in constant increase all over the world and affects 35% of the global population according to the World Health Organisation. It is associated with other cardiovascular risk factors (particularly hypertension and diabetes) and with high morbi-mortality. It is also responsible for an increase of the risk of developing chronic kidney diseases (CKD). In fact, obese patients represent 25% of the dialysis population and Picardy is one of the most affected areas. However, their access to kidney transplant is still restricted and the reasons are not completely understood.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old.
* Patients with BMI≥30 kg/m2 (for study population) and 25≤BMI≤30 kg/m2(for control population) one month after dialysis initiation.
* Patients agree with their data collection.

Exclusion Criteria:

* Patients with bariatric surgery history.
* Patients needed dialysis for graft dysfunction.
* Data loss.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will be included in the study one month after the dialysis initiation. All clinical (obesity history, comorbidities, nephropathy aetiology and treatment…) and biological (nutrition markers, hemoglobin, brain natriuretic peptide (BNP)…) informations after one month and during the two years of follow-up (weight evolution, obesity complications, transplant path...) will be collected.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-03-16 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
variation of pre-transplant status two years after the obese patients' dialysis initiation between both groups | two years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No